CLINICAL TRIAL: NCT04293224
Title: Metabolic and Bio-behavioral Effects of Following Recommendations in the Dietary Guidelines for Americans
Acronym: DGA4ME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FL111
Record Dates: First submitted 2020-02-27; First posted 2020-03-03 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Body Weight
Keywords: Dietary Guidelines for Americans; Physical Activity for Americans; Mediterranean Diet; Controlled Feeding; Women; PreDiabetes; Metabolic Syndrome; Cognitive Function; Stress, Physiological; Executive Function; Cardiovascular Diseases; Cardiovascular Risk Factor; Eating Behavior; Glucose Intolerance; Metabolomic Profiling; Metabolic flexibility; Gut Microbiome; Genome Testing; Prehypertension; Insulin Resistance; Insulin Sensitivity; Hypertriglyceridemic; Waist to Hip Ratio; Allostatic Load; Physiology
MeSH Terms: conditions — Obesity; Body Weight; Prediabetic State; Metabolic Syndrome; Cardiovascular Diseases; Feeding Behavior; Glucose Intolerance; Prehypertension; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DGA Mediterranean diet pattern, energy balance (Experimental): Diet plan focused on energy balance (meets calorie needs), emphasizes fruits, vegetables and whole grains and limits calories from added sugars and saturated fats and reduces sodium intake per Dietary Guidelines for Americans (DGA) recommendations.
  Interventions: Other: DGA Mediterranean diet pattern, energy balance
- DGA Mediterranean diet pattern, negative energy balance (Experimental): Negative energy balance (~25% calorie reduction compared to needs), emphasizes fruits, vegetables and whole grains and limits calories from added sugars and saturated fats and reduces sodium intake per Dietary Guidelines for Americans (DGA) recommendations.
  Interventions: Other: DGA Mediterranean diet pattern, negative energy balance
- TAD diet pattern (Experimental): Typical American Diet (TAD) with negative energy balance (~25% calorie reduction compared to needs) which mimics intake of fruits, vegetables, whole grains, added sugars, saturated fats and sodium based on data from What We Eat in America (WWEIA).
  Interventions: Other: TAD diet pattern, negative energy balance

INTERVENTIONS:
Other: DGA Mediterranean diet pattern, energy balance — Foods and beverages will be provided for participants for eight weeks. During the controlled feeding portion of the study the DGA Mediterranean diet pattern will be based on the Table A7-1 of the 2015 Dietary Guidelines for Americans which outlines daily nutritional goals for age-sex groups based on Dietary Reference Intakes (DRI) and dietary guidelines recommendations.
  Arms: DGA Mediterranean diet pattern, energy balance
Other: DGA Mediterranean diet pattern, negative energy balance — Foods and beverages will be provided for participants for eight weeks. During the controlled feeding portion of the study the DGA Mediterranean diet pattern will be based on the Table A7-1 of the 2015 Dietary Guidelines for Americans which outlines daily nutritional goals for age-sex groups based on Dietary Reference Intakes (DRI) and dietary guidelines recommendations
  Arms: DGA Mediterranean diet pattern, negative energy balance
Other: TAD diet pattern, negative energy balance — Foods and beverages will be provided for participants for eight weeks. During the controlled feeding portion of the study the be based on evidence collected from What We Eat in America (WWEIA) data. Based on this data the participants will be provided a diet that reflects American dietary trends.
  Arms: TAD diet pattern

SUMMARY:
This study, at the Western Human Nutrition Research Center (WHNRC), will focus on whether or not achieving and maintaining a healthy body weight is the most important health promoting recommendation of the Dietary Guidelines for Americans (DGA).The investigators hypothesize that improvement in cardiometabolic risk factors resulting from eating a DGA style diet will be greater in people whose energy intake is restricted to result in weight loss compared to those who maintain their weight. The investigators further propose that during a state of energy restriction, a higher nutrient quality diet such as the DGA style diet pattern, will result in greater improvement in cardiometabolic risk factors compared to a typical American diet (TAD) pattern that tends to be lower nutrient quality (more energy-dense and less nutrient-rich.)

DETAILED DESCRIPTION:
This will be a 28-week study including pre-diet testing (week 1), an 8-week controlled feeding period, post-diet testing (week 10), a follow-up period of dietary education and observation, and end of study testing (week 28). During the 8 week feeding, participants will be randomly assigned one of the following diets:

1. DGA Mediterranean diet pattern at sufficient energy level to maintain body weight (energy balance)
2. DGA Mediterranean diet pattern at a moderately reduced energy level (negative energy balance)
3. TAD diet pattern at a moderately reduced energy level (negative energy balance)

In the follow-up phase, the investigators will evaluate how multiple factors may influence body weight management, including previous dietary exposure, as well as the role of cognitive function, executive function, genetics, habitual diet, physical activity, eating behavior, stress and stress responsivity, metabolic flexibility and gut microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) 23-39.9 kg/m2 or 32-50% body fat percentage
* Willingness to have blood drawn
* The criteria listed above and at least one of the following: Fasting glucose ≥100 mg/dL but <126 mg/dL or Fasting triglyceride ≥125 mg/dL or HDL-cholesterol ≤50 mg/dL or Blood Pressure (BP): Systolic BP ≥130 mmHg or Diastolic BP ≥85 mmHg or Hemoglobin A1C ≥ 5.7 and <6.5%

Exclusion Criteria:

* Active participation in another research study
* Tested positive for COVID-19 within the past 10 days
* Been in close contact with a COVID-19 positive person within the past 14 days
* Blood Pressure (BP): Systolic BP ≥140 mmHg or Diastolic BP ≥90 mmHg
* LDL cholesterol ≥190 mg/dL
* Triglycerides ≥500 mg/dL
* Current use of smoking or chewing tobacco, e-cigarettes, cigars, vaping, cannabis or other use of nicotine containing products (within the past 6 months)
* Current use of dietary supplements and/or unwillingness to cease intake of dietary supplements
* Vegan or vegetarian lifestyle or any other dietary restrictions that would interfere with consuming the intervention foods and beverages (including dietary intolerances, allergies and sensitivities)
* Unwillingness to consume intervention foods and beverages
* Engage in more than moderate drinking (> 1 drink serving per day) or binge drinking (4 drinks within two hours).
* Unwillingness to cease alcohol intake as required for specific duration of the study
* Excessive intake of caffeine containing products (excessive defined as ≥ 400 mg/day)
* Unwillingness to refrain from caffeine intake on lab visit days.
* Intentional weight change of ≥5% of body weight within 6 months of entry into the study
* Diagnosis of disordered eating or eating disorder
* Recent diagnosis of any of the following or measurement on screening lab tests: Anemia (hemoglobin <11.7 g/dL) or abnormal liver or thyroid function (defined as liver enzymes that are >200% of upper limit (ALT upper limit is 43 U/L or Aspartate transaminase (AST) upper limit is 54 U/L) and thyroid function tests: Thyroxine (T4, free) <0.56 or >1.64 ng/dL; Thyroid-stimulating hormone (TSH) <0.35 or >5.6 μIU/mL).
* History of any of the following: Gastric bypass surgery, inflammatory bowel disease (IBD) or other GI conditions that would interfere with consuming the intervention foods, active cancer in the past three years excluding squamous or basal cell carcinomas of the skin that have been handled medically by local excision and other serious medical conditions
* Recent dental work or have conditions of the oral cavity that would interfere with consuming the intervention foods and beverages
* Taking any medication in the class of antipsychotics
* Long term use of antibiotics
* Taking any over the counter or prescribed medication for any of the following: Elevated lipids, elevated glucose, high blood pressure, weight loss or conditions that require corticosteroids (e.g. asthma, arthritis or eczema).
* Are pregnant, planning to become pregnant within the duration of the study or breastfeeding.

Ages: 19 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in body weight | Measured weekly for weeks 1 through 10, and weeks 13, 17, 21, 24 and 28
  Body weight will be measured to the nearest 0.1 kg using a calibrated electronic scale.

SECONDARY OUTCOMES:
Height | Week 1
  Height will be measured to the nearest 0.1 cm using a wall-mounted stadiometer.
Change in body mass index | Measured weekly for weeks 1 through 10, and weeks 13, 17, 21, 24 and 28
  Body weight and height will be used to calculate Body Mass Index (BMI) as kg/m2.
Change in body water (via InBody) | Week 1, 10, 28
  Measured using bioelectrical impedance analysis (BIA) with an InBody 770® expressed as kg.
Change in body fat (via DEXA scan) | Week 1, 10, 28
  Fat mass (grams) will be measured using dual energy x-ray absorptiometry (DEXA).
Change in waist circumference | Week 1, 10, 28
  Waist circumference is measured with an anthropometric tape. Measurements will be performed in duplicate and averages recorded to the nearest 0.1 cm.
Change in hip circumference | Week 1, 10, 28
  Hip circumference is measured with an anthropometric tape. Measurements will be performed in duplicate and averages recorded to the nearest 0.1 cm.
Change in waist to hip ratio | Week 1, 10, 28
  Waist and hip circumference will be expressed as a ratio.
Change in resting systolic blood pressure | Week 1, 10, 28
  Blood pressure will obtained via automated instrument and blood pressure cuff. At least two measurements will be made, expressed in mmHg, and the average value will be recorded.
Change in resting diastolic blood pressure | Week 1, 10, 28
  Blood pressure will obtained via automated instrument and blood pressure cuff. At least two measurements will be made, expressed in mmHg, and the average value will be recorded.
Change in resting heart rate | Week 1, 10, 28
  Resting heart rate (pulse) will obtained via automated instrument in beats per minute.
Genetic Risk of Obesity | Week 1
  Genomic DNA will be collected from white blood cells. A polygenic risk score (PRS) indexing genetic predisposition to obesity using known obesity single nucleotide polymorphisms (SNPs).
Change in vascular health | Week 1, 5, 10
  Peripheral Arterial Tone (PAT) technology will be used to measure vascular health. The EndoPAT test is a non-invasive measurement of the overall health of the endothelium.
Change in liver fat | Week 1 and 10
  Liver fat assessed from the Controlled Attenuation Parameter (CAP) computed from the liver stiffness measurement using the Fibroscan®
Change in liver stiffness | Week 1 and 10
  Liver stiffness assessed from the shear wave speed with pulse echo ultrasound using the Fibroscan®
Change in blood metabolite profiles | Week 1 and 10
  Analysis of metabolites, the small molecule substrates, intermediates and products of metabolism analyzed by mass spectrometry (MS). Includes branched chain amino acids, 2 hydroxybutyric acid, acylcarnitines, saturated, monounsaturated and polyunsaturated non-esterified fatty acids, triglyceride species, phospholipid species, bile acids and steroid hormones.
Change in fasting blood glucose | Week 1, 10, 28
  This outcome will evaluate blood sugars levels in the fasted state.
Change in hemoglobin A1C | Week 1, 10, 28
  This outcome will evaluate glycated hemoglobin as a reflection of the plasma glucose level during the past two to three months.
Change in urinary sodium | Week 1, 5, 7 and 10
  Urinary sodium will be measured as indicators of dietary compliance during the feeding intervention of the study. All urine passed for a 24 hour period will be collected.
Change in urinary potassium | Week 1, 5, 7 and 10
  Urinary potassium will be measured as indicators of dietary compliance during the feeding intervention of the study. All urine passed for a 24 hour period will be collected.
Change in urinary nitrogen | Week 1, 5, 7 and 10
  Urinary nitrogen will be measured as indicators of dietary compliance during the feeding intervention of the study. All urine passed for a 24 hour period will be collected.
Change in red blood cell fatty acids | Week 1, 10, 28
  Red blood cell fatty acids will be analyzed by mass spectrometry (MS).
Change in C-reactive protein | Week 1, 10, 28
  C-Reactive Protein will be measured as a non-specific marker for inflammation.
Change in carotenoid levels | Week 1 and 10
  Serum carotenoids, including vitamin A, alpha-carotene, and beta-carotene will be used to evaluate nutrient status and dietary intake of vegetables prior to feeding intervention and post feeding intervention.
Change in total cholesterol | Week 1 and 10
  Total cholesterol will be collected to evaluate cardiac risk expressed as milligrams per deciliter (mg/dL).
Change in high density lipoprotein (HDL) cholesterol | Week 1 and 10
  HDL cholesterol will be collected to evaluate cardiac risk expressed as milligrams per deciliter (mg/dL).
Change in low density lipoprotein (LDL) cholesterol | Week 1 and 10
  LDL cholesterol will be collected to evaluate cardiac risk expressed as milligrams per deciliter (mg/dL).
Change in triglycerides in response to a meal | Baseline and 1, 2, 3, and 6 hours after a challenge meal
  Triglycerides will be measured in blood (mg/dL).
Change in ghrelin in response to a meal | Baseline and 1, 2, 3, and 6 hours after a challenge meal
  Ghrelin will be evaluated as an indicator of hunger signaling.
Change in leptin in response to a meal | Baseline and 1, 2, 3, and 6 hours after a challenge meal
  Leptin will be evaluated as an indicator of satiety signaling.
Change in insulin in response to a meal | Baseline and 1, 2, 3, and 6 hours after a challenge meal
  Insulin measured in blood using an antibody based assay. Will also be expressed as the quantitative insulin sensitivity check index (QUICKI).
Change in Matsuda Index | Baseline and 1, 2 hours after a challenge meal
  Matsuda index will be calculated from plasma glucose and insulin.
Change in resting metabolic rate | Week 1 and 10
  Respiratory gas exchange measurements (oxygen consumption-VO2 and carbon dioxide production-VCO2) will be made to determine metabolic rate using a metabolic cart system.
Change in post-prandial metabolic rate | 1, 2, 3 and 6 hours after a meal
  Post-prandial metabolic rate measured using indirect calorimetry.
Change in metabolic flexibility | Week 1 and 10
  The formula is designed to deliver approximately 800 kcals total with 60% kcals from fat (approximately 55 g of fat), 25% kcals from carbohydrates, and 15% of kcals from protein.
Change in predicted VO2 max | Week 1, 10, 28
  Cardiorespiratory endurance will be evaluated by measuring heart rate (HR) and oxygen consumption (VO2) during a walking graded exercise test on a treadmill.
Change in interstitial glucose levels | Week 1 and 10
  A continuous glucose monitor (CGM) will be used to continuously assess interstitial glucose levels. The Abbott Freestyle Libre Pro Sensor is inserted under the skin on the back of the arm. The sensor will measure the interstitial glucose level every fifteen minutes. Participants will wear the monitors for fourteen days.
Change in executive function | Week 1 and 10
  Assessed using Cambridge Gambling Task (CGT), from Cambridge Neuropsychological Test Automated Battery (CANTAB).
Change in response speed | Week 1 and 10
  Assessed using Motor Screening Task (MOT), from Cambridge Neuropsychological Test Automated Battery (CANTAB).
Change in verbal memory | Week 1 and 10
  Assessed using Verbal Recognition Memory (VRM) task from Cambridge Neuropsychological Test Automated Battery (CANTAB).
Change in psycho-motor speed | Week 1 and 10
  Assessed using Reaction Time (RTI) task from Cambridge Neuropsychological Test Automated Battery (CANTAB).
Change in spatial memory | Week 1 and 10
  Assessed using Spatial Working Memory (SWM) task from Cambridge Neuropsychological Test Automated Battery (CANTAB).
Change in multitasking | Week 1 and 10
  Assessed using Multitasking Test (MTT) from Cambridge Neuropsychological Test Automated Battery (CANTAB).
Change in social cognition | Week 1 and 10
  Assessed using Emotional Recognition (ERT) task from Cambridge Neuropsychological Test Automated Battery (CANTAB).
Change in attentive function | Week 1 and 10
  Assessed using Stop Signal Task (STT) from Cambridge Neuropsychological Test Automated Battery (CANTAB).
Change in allostatic load | Week 1, 10, 28
  Allostatic load (AL) is an aggregate value derived from several parameters that assess physiologic adaptive response to neural or neuroendocrine stressors. The following measures are used to determine the AL score: Urinary cortisol and catecholamine levels, resting blood pressure, waist to hip ratio, blood levels of high sensitivity C-Reactive Protein, cholesterol, dehydroepiandrosterone sulfate and hemoglobin A1c, and urinary levels of epinephrine and norepinephrine.
Change in continuous systolic blood pressure | Week 1 and 10
  Blood pressure measured using a Continuous Non-invasive Arterial Pressure (CNAP®) device in mmHg.
Change in continuous diastolic blood pressure | Week 1 and 10
  Blood pressure measured using a Continuous Non-invasive Arterial Pressure (CNAP®) device in mmHg.
Change in mean arterial blood pressure | Week 1 and 10
  Blood pressure measured using a Continuous Non-invasive Arterial Pressure (CNAP®) device in mmHg .
Change in mood | Week 1 and 10
  Mood assessed using the Profile of Mood States (POMS). Total Mood Disturbance (TMD) score is found from the difference between "negative" subscales - "positive" subscales. Individual scores on the POMS range from -32 to 200 with higher scores indicating higher mood disturbance.
Change in perceived stress | Week 1, 6, 10, 19 and 28
  Perceived stress measured using the Perceived stress scale (PSS). Scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress. Responses for individual questions are summed to a total score.
Change in self-efficacy | Week 10, 19 and 28
  This 20 item questionnaire is a measurement of the capacity to execute behaviors necessary to change their weight and begin to implement exercise in their lives regularly.
Change in diet satisfaction | Week 1, 19 and 28
  This 28 item questionnaire acts as a valid instrument for assessing diet satisfaction in the context of weight-management. This measurement assesses diet satisfaction both within and outside the context of weight-loss treatment, as well as to assesses change in satisfaction as a result of treatment.
Change in appetite | Week 1 and 10
  A computer tablet with stylus will be used to assess hunger and appetite, defined as perceived hunger, fullness, desire to eat, prospective consumption and other measures of food craving and perceived hypoglycemia. Questions will be presented one-by-one on the screen and participants will be asked to express their response using visual analog scales (VAS). This measurement will be evaluated during the meal challenge assessment.
Three factor eating questionnaire | Week 1 and 10
  This 18 item questionnaire is used to examine three dimensions of human eating behavior including cognitive restraint, disinhibition or uncontrolled eating and hunger.
Barriers to physical activity | Week 1
  Participants will be asked to complete the Barriers to Being Active questionnaire.
Usual physical activity | Week 1
  An accelerometer (Actical) will be continuously worn by participants during waking hours (excluding bathing and swimming) for a period of 7 days.The measure of usual physical activity is used to estimate total energy expenditure and energy requirements.
Diet acceptability | Week 10
  This measurement is an evaluation of palatability, ease of preparation, satisfaction, and perceived benefits and adverse effects related to a prescribed controlled feeding diet.
Yale Food Addiction Scale | Week 1
  Measures markers of substance dependence with the consumption of high fat/high sugar foods. This is a 25-item self-report measure that includes mixed response categories (dichotomous and Likert-type format).
Changes in dietary intake | Week 1, 19, and 28
  Three non-consecutive twenty-four hour dietary recalls will be collected when subjects are self-selecting their 'usual' diets. A three day average nutrient intake will be expressed.
Change in stress reactivity | Week 1 and 10
  Acute stress reactivity will be assessed by measuring salivary cortisol concentrations in response to a challenging task.
Change in heart rate variability | Week 1 and 10
  Autonomic physiological functioning will be assessed using the MindWare Cardio/Galvanic Skin Response (GSR) system, a device that connects to the subject's torso with eight disposable electrodes and a heart rate monitor. Emotional arousal via skin conductance, a form of electrodermal activity (EDA) is also measured.
Change in Food Choice | Week 1 and 10
  Food choice computer-based tests from Leeds, United Kingdom, will be used to estimate explicit liking and implicit wanting for several different categories of foods.
Change in oxygen consumption rate (OCR) | Week 1 and 10
  Measured in peripheral blood mononuclear cells by use of Seahorse XF Analyzer, a tool for measuring glycolysis and oxidative phosphorylation (through oxygen consumption) simultaneously in the same cells.
Change in extracellular acidification rate (ECAR) | Week 1 and 10
  Measured in peripheral blood mononuclear cells by use of Seahorse XF Analyzer, a tool for measuring glycolysis and oxidative phosphorylation (through oxygen consumption) simultaneously in the same cells.
Change in fecal microbiome | Week 1, 10 an 28
  Assays will be performed on fecal samples to determine DNA representing the colonic microbiota.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin D Laugero, PhD, Principal Investigator — USDA, Western Human Nutrition Research Center
Locations (1):
- UC Davis, Western Human Nutrition Research Center, Davis, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized metabolomics data will be deposited on Metabolomics Work Bench (https://www.metabolomicsworkbench.org/), a national and international repository for metabolomics data and metadata, developed in support of the National Institutes of Health (NIH) Common Fund Metabolomics Program and housed at the San Diego Supercomputer Center (SDSC), University of California, San Diego. Archived data will include raw data files, quality assurance data, final analytical data, and associated experimental metadata including experimental group assignments, anthropometric, physiological and clinical measures.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data.

REFERENCES:
- [Background] Krishnan S, Adams SH, Allen LH, Laugero KD, Newman JW, Stephensen CB, Burnett DJ, Witbracht M, Welch LC, Que ES, Keim NL. A randomized controlled-feeding trial based on the Dietary Guidelines for Americans on cardiometabolic health indexes. Am J Clin Nutr. 2018 Aug 1;108(2):266-278. doi: 10.1093/ajcn/nqy113. PMID 30101333
- See also: WHNRC website — https://www.ars.usda.gov/pacific-west-area/davis-ca/whnrc/